CLINICAL TRIAL: NCT01360268
Title: The Metabolic Profile and Adipocytokine Alterations of Patients With HCV Infection Before and After HCV Therapy"
Brief Title: The Metabolic Profile and Adipocytokine Alterations of Patients With HCV Infection Before and After HCV Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Ming-Ling Chang/ M.D., Liver Research Unit,Division of Hepatology, Department of Hepatogastroenterology,Chang Gung memorial Hospital, Taoyuan, Taiwan
Other Study IDs: Merck (MISP) # 38846
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-02

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale for this study:

Correction of hypocholesteremia and insulin resistance after successful eradication of HCV by combination therapy of interferon and ribavirin has been shown in several studies. The majority of these studies examined genotype 1 and some genotype 3 patients, but it is not clear if the same results can be achieved in other genotypes of HCV.

Moreover, clinical data of the relationships between different adipocytokines, metabolic profiles, and HCV and treatment is of value to further understand the mechanisms for HCVrelated metabolic alterations. The present proposal is designed to address the paradox of HCV-related metabolic alterations/adipocytokine alterations and to determine how BMI influences the HCV-related metabolic alteration/adipocytokine aterations by collecting and analyzing the samples from humans with HCV infection prior to and after combination of peginterferon alpha-2b plus ribavirin

For metabolic alternations:

Lipid profile: After treatment, responders in both genotype I and II will experience more increase of cholesterol levels and LDL levels than nonresponders/ relapseres. Insulin resistance: After treatment, responders with both genotype I and II will experience more decrease of HOMA-IR than nonresponders/ relapseres; higher percentage of responders will achieve HOMA-IR < 2 than nonresponders/ relapseres B. For adipocytokine alternation, this study is more of exploratory propose as there is still little well established consensus.

DETAILED DESCRIPTION:
Subjects with chronic hepatitis C infections will be enrolled

Inclusion Criteria

1. Aged 18 y/o or older
2. Positive for the HCV antibody and HCV RNA detected
3. Patients with abnormal liver function OR a liver biopsy specimen taken in the 6 months prior to study entry showing chronic hepatitis, or liver fibrosis, or liver cihhrosis
4. Have not been previously treated with pegylated-interferon and ribavirin for HCV
5. Genotype 1 or Genotype 2

Exclusion Criteria

1. Subjects with decompensated liver disease
2. With human immunodeficiency virus
3. With hepatitis B infection
4. With hemochromatosis defined by a pre-existing diagnosis of hemochromatosis or a positive HFE gene mutation or recipients of solid organ transplants
5. With clinically significant cardiac or cardiovascular abnormalities, organ grafts, systemic infections, clinically significant bleeding disorders, evidence of malignant neoplastic diseases
6. Subjects who are on lipid-lowering medications
7. Poorly controlled Diabetes (A1C > 9%) The study will go through the CGMH IRB review and be posted into clinicaltrial.gov.

This is a single centre, prospective, open-label, single arm, interventional study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 y/o or older
2. Positive for the HCV antibody and HCV RNA detected
3. Patients with abnormal liver function OR a liver biopsy specimen taken in the 6 months prior to study entry showing chronic hepatitis, or liver fibrosis, or liver cihhrosis
4. Have not been previously treated with pegylated-interferon and ribavirin for HCV
5. Genotype 1 or Genotype 2

Exclusion Criteria:

1. Subjects with decompensated liver disease
2. With human immunodeficiency virus
3. With hepatitis B infection
4. With hemochromatosis defined by a pre-existing diagnosis of hemochromatosis or a positive HFE gene mutation or recipients of solid organ transplants
5. With clinically significant cardiac or cardiovascular abnormalities, organ grafts, systemic infections, clinically significant bleeding disorders, evidence of malignant neoplastic diseases
6. Subjects who are on lipid-lowering medications
7. Poorly controlled Diabetes (A1C > 9%) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic hepatitis C infections
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Ling Chang, Principal Investigator — CGMH
Locations (1):
- Ming-Ling Chang, Dawan, Taiwan, Taiwan